CLINICAL TRIAL: NCT02759432
Title: Effect of a 4-week Fun Fast Interval Training (FFIT) Activity Programme on Physical Fitness and Quality of Life in Adolescent School Pupils
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teesside University (Other)
Responsible Party: Principal Investigator, Kathryn Weston, Dr, Teesside University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TEES-046/16
Record Dates: First submitted 2016-04-29; First posted 2016-05-03 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: High-intensity Interval Training
Keywords: high-intensity interval training; adolescents; physical fitness; quality of life; school-based intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Participants in the intervention group will complete a 4-week school-based high-intensity interval exercise training programme. The intervention will take place twice per week, and comprise of 6-8 repetitions of 45 s maximal effort exercise (boxing, running, soccer and basketball drills), each interspersed with 90-s rest. Participants will be encouraged to work maximally during the 45-s repetitions.
  Interventions: Other: High-intensity interval exercise training
- Control (No Intervention): Participants in the control group will be instructed not to change their lifestyle, dietary or physical activity habits during the intervention period, and maintain their normal school physical education routine

INTERVENTIONS:
Other: High-intensity interval exercise training
  Arms: Intervention

SUMMARY:
Low-volume high-intensity interval exercise training may improve aspects of health and fitness in young people, but the effect of this type of exercise on quality of life has yet to be assessed. The investigators aim to examine the effect of a 4-week school-based low-volume high-intensity interval training programme (called the Fun Fast Interval Training [FFIT] activity project) on physical fitness and quality of life in adolescent school pupils. Approximately 145 English adolescents aged 11-12 years will be approached and invited to take part in the study. Participants will be healthy female volunteers, recruited from one school in Northeast England. Using a non-randomised design, one school year group will be assigned to take part in the intervention, and a second year group assigned to the control condition.Those in the intervention group will complete a 4-week school-based high-intensity interval exercise training programme. The intervention will take place twice per week, and comprise of 6-8 repetitions of 45 s maximal effort exercise (boxing, running, soccer and basketball drills), each interspersed with 90-s rest. Participants will be encouraged to work maximally during the 45-s repetitions. Control participants will be instructed not to change their lifestyle, dietary or physical activity habits during the intervention period, and maintain their normal school physical education routine. Study outcomes will be 20 m shuttle run test performance, health-related quality of life, standing broad jump performance, hand dynamometer performance, waist circumference and 10 m and 20 m sprint performance.

ELIGIBILITY:
Inclusion Criteria:

1. Must be in school Year 7 or 8 at the school where the study will take place
2. Must provide parental consent and participant assent
3. Must be free from exclusion criteria

Exclusion Criteria:

1. Symptoms of or known presence of heart disease or major atherosclerotic cardiovascular disease.
2. Condition or injury or co-morbidity affecting the ability to undertake exercise.
3. Diabetes mellitus
4. Early family history of sudden death
5. Pregnancy or likelihood of pregnancy

Ages: 11 Years to 13 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 132 (Actual)
Dates: Start 2016-05; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline (0 weeks) cardiorespiratory fitness (assessed via the 20 m shuttle run test performance test) at the post-intervention time point (4 weeks) | Baseline (0 weeks) and post-intervention (4 weeks)
  Cardiorespiratory fitness will be indirectly assessed by participants performing the 20 m shuttle run test. Test performance is expressed in number of shuttle completed
Change from baseline (0 weeks) leg power (assessed via standing broad jump performance at the post-intervention time point (4 weeks) | Baseline (0 weeks) and post-intervention (4 weeks)
  Leg power will be assessed by participants performing a standing broad jump test. Test performance is expressed as distance jumped.
Change from baseline (0 weeks) upper body strength (assessed via handgrip dynamometer performance) at the post-intervention time point (4 weeks) | Baseline (0 weeks) and post-intervention (4 weeks)
  Upper body strength will be assessed by participants performing the handgrip dynamometer test. Test performance is expressed as grip strength measured in kilogrammes.
Change from baseline (0 weeks) in 10 m running speed (assessed via 10 m sprint performance at) the post-intervention time point (4 weeks) | Baseline (0 weeks) and post-intervention (4 weeks)
  10 m running speed will be assessed by participants completing a 10 m running sprint. Test performance is expressed in seconds.
Change from baseline (0 weeks) in 20 m running speed (assessed via 20 m sprint performance at) the post-intervention time point (4 weeks) | Baseline (0 weeks) and post-intervention (4 weeks)
  20 m running speed will be assessed by participants completing a 20 m running sprint. Test performance is expressed in seconds.
Change from baseline (0 weeks) waist circumference at the post-intervention time point (4 weeks) | Baseline (0 weeks) and post-intervention (4 weeks)
  Measurements will be expressed in centimetres.
Change from baseline (0 weeks) health-related quality of life (assessed via completion of the Kid-Kindl questionnaire [Ravens-Sieberer & Bullinger, 2000] at the post-intervention time point (4 weeks) | Baseline (0 weeks) and post-intervention (4 weeks)

OTHER OUTCOMES:
Heart rate during high-intensity interval exercise training sessions | Up to 4 weeks
Rating of perceived exertion (assessed via the Children's scale of perceived exertion [Robertson et al., 2000) during high intensity interval exercise training sessions | Up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn L Weston, PhD, Principal Investigator — Teesside University, Middlesbrough, UK
Locations (1):
- Outwood Academy Ormesby, Middlesbrough, United Kingdom